CLINICAL TRIAL: NCT05134116
Title: Cerebral Near-infrared Spectroscopy Monitoring Versus Treatment as Usual for Extremely Preterm Infants: a Protocol for the Follow-up Study for the SafeBoosC-III Trial
Brief Title: SafeBoosC III Two-year Follow-up
Status: Completed | Type: Observational
Sponsor: Gorm Greisen (Other)
Responsible Party: Sponsor-Investigator, Gorm Greisen, Professor, Cheif Consultant Neonatologist, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Other Study IDs: SafeBoosC-IIIfu
Record Dates: First submitted 2021-10-19; First posted 2021-11-24 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Deficits, Neurologic; Extreme Prematurity; Brain Damage
Keywords: Neurodevelopmental disability; Cerebral palsy; Neurosensory deficits; Cognitive disability; Follow up study; Extremely preterm birth; Near infrared spectroscopy (NIRS); Cerebral oximetry
MeSH Terms: conditions — Neurologic Manifestations; Brain Injuries; Cerebral Palsy | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Treatment as usual + cerebral oximetry monitoring the first 72 hours of life — SafeBoosC - Safeguarding the Brain of Our Smallest Children - an Investigator-initiated Randomised, Blinded, Multinational, Phase II Feasibility Clinical Trial on Near-infrared Spectroscopy Monitoring Combined With Defined Treatment Guidelines Versus Standard Monitoring and Treatment as Usual in Premature Infants

SUMMARY:
The SafeBoosC-III 2 year follow up study will follow up on all patients randomised in the SafeBoosC-III clinical trial (NCT03770741). The investigators will collect data when the patients are two years of corrected age from routine standardised follow up assessments, parental questionnaires as well as informal assessments. The study will commence in September 2021, and will expect to include all 72 sites across 18 countries, which take part of the SafeBoosC-III clinical trial.

DETAILED DESCRIPTION:
In the SafeBoosC-III trial, the objective is to investigate the effect of treatment based on cerebral near-infrared spectroscopy (NIRS) monitoring of brain oxygenation compared with treatment as usual in extremely preterm infants. The primary outcome of the trial is death or survival with severe brain injury at 36 weeks' postmenstrual age. Despite an association between severe brain injury diagnosed in the neonatal period and later neurodevelopmental disability, this relationship is not always strong. Therefore, if treatment based on cerebral NIRS monitoring decreases the risks of death or survival with severe brain injury, it is important to document if the beneficial effect persists into early childhood, in the form of better neurodevelopmental outcome. Furthermore, it is also important to identify evidence of unexpected harms. It would be unfortunate if cerebral NIRS monitoring became standard practice without good evidence that long-term patient-relevant benefits outweigh possible harms. As the SafeBoosC-III trial intends to randomise 1600 infants, there is potential to achieve sufficient power for a meaningful assessment of the experimental intervention's effect on long-term neurodevelopment, as well as an evaluation of unexpected harms. The objective of the SafeBoosC III follow-up study is to investigate the benefits and harms of treatment guided by cerebral NIRS monitoring of brain oxygenation in extremely preterm infants during the first 72 hours of life, assessed at two years' corrected age. The hypothesis is that the intervention will decrease a composite of death or moderate-or-severe neurodevelopmental disability at two years' corrected age, and/or increase cognitive function in survivors assessed by the Bayley III/IV test, with insignificant harms. The investigators aim to collect data on as many children as possible and will do this by collecting clinical data from health care records as well as answers from parental questionnaires.

ELIGIBILITY:
Inclusion Criteria:

Participation in the SafeBoosC-III trial and enrollment in a neonatal intensive care unit (NICU) taking part in the follow-up study, with parental consent according to local regulations.

Exclusion Criteria:

Parental objection to the use of their child's data in the follow-up study.

Ages: 12 Months to 30 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants born below 28 weeks of gestation and randomised in the SafeBoosC-III trial
Sampling Method: Non-Probability Sample
Enrollment: 1601 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2024-10-19 (Actual); Study Completion 2024-10-19 (Actual)

PRIMARY OUTCOMES:
Death or moderate-or-severe neurodevelopmental disability | To be assessed at two years of corrected age
  A child will be classified with moderate-or-severe neurodevelopmental disability if they have been diagnosed with cerebral palsy, a cognitive function score below -2 standard deviations from the norm, hearing impairment, or vision impairment or from data from a parental questionnaire.
Mean Bayley III/IV cognitive score | To be assessed at two years of corrected age
  The cognitive scores from the Bayley III/IV assessment will constitute a single continuous outcome measure (higher scores meaning better outcomes)

OTHER OUTCOMES:
Daily medication the last two months (yes/no) | To be assessed at two years of corrected age
  Will be assessed based on the childs health care records or a parental questionnaire
Any other chronic illness (defined as any problem which has been diagnosed by a doctor and which 1) is expected to last more than a few months, 2) causes problems in everyday life, or 3) is a risk of early death or disability), | To be assessed at two years of corrected age
  Will be assessed based on the childs health care records or a parental questionnaire
Growth measurements | To be assessed at two years of corrected age
  Mean head circumference, mean height and mean body weight. Will be assessed based on the childs health care records
Components of the co-primary outcomes | To be assessed at two years of corrected age
  All components of the co-primary outcomes will be reported for the two groups separately as well as effect estimates with confidence intervals and will be taken into consideration when interpreting the main results

CONTACTS AND LOCATIONS:
Locations (1):
- Righospitalet (The University Hospital, Copenhagen), Copenhagen, Denmark

REFERENCES:
- [Derived] Rasmussen MIS, Hansen ML, Pellicer A, Gluud C, Dempsey E, Mintzer J, Hyttel-Sorensen S, Heuchan AM, Hagmann C, Ergenekon E, Dimitriou G, Pichler G, Naulaers G, Tkaczyk J, Fuchs H, Fumagalli M, Nesargi S, Fredly S, Szczapa T, Plomgaard AM, Hansen BM, Olsen MH, Jakobsen JC, Greisen G. Cerebral oximetry monitoring versus usual care for extremely preterm infants: a detailed statistical analysis plan for the 2-year follow-up of the participants of the SafeBoosC-III randomised clinical trial. Trials. 2026 Jan 5. doi: 10.1186/s13063-025-09392-7. Online ahead of print. PMID 41491571
- [Derived] Rasmussen MI, Hansen ML, Pellicer A, Gluud C, Dempsey E, Mintzer J, Hyttel-Sorensen S, Heuchan AM, Hagmann C, Ergenekon E, Dimitriou G, Pichler G, Naulaers G, Cheng G, Tkaczyk J, Fuchs H, Fumagalli M, Nesargi S, Fredly S, Szczapa T, Plomgaard AM, Hansen BM, Jakobsen JC, Greisen G. Cerebral oximetry monitoring versus usual care for extremely preterm infants: a study protocol for the 2-year follow-up of the SafeBoosC-III randomised clinical trial. Trials. 2023 Oct 7;24(1):653. doi: 10.1186/s13063-023-07653-x. PMID 37805539
- See also: Trial and Follow up website — http://safeboosc.eu

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/16/NCT05134116/Prot_SAP_000.pdf